CLINICAL TRIAL: NCT01352663
Title: An Open Label, Randomized Comparison of Wockhardt's Recombinant Insulin Analogue With Innovator's Glargine in Type 1 Diabetic Patients.
Brief Title: Immunogenicity Safety Study of Wockhardt's Recombinant Insulin Analogue in Type 1 Diabetic Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business strategy decision
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P3-GLR-IMSFDA-01
Record Dates: First submitted 2011-05-09; First posted 2011-05-12 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Type I Diabetes
Keywords: Type I Diabetes; Wockhardt; Insulin Analogue
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wockhardt's Insulin Analogue (Recomb) (Experimental): Basal bolus Wockhardt's Recombinant Insulin Analogue to be injected subcutaneously.
  Interventions: Biological: Wockhardt's Insulin Analogue (Recomb)
- Lantus® (Active Comparator): Basal bolus Insulin analog glargine (Lantus®) to be injected subcutaneously.
  Interventions: Biological: Lantus®

INTERVENTIONS:
Biological: Wockhardt's Insulin Analogue (Recomb) — Basal bolus Wockhardt's Recombinant Insulin Analogue to be injected subcutaneously.
  Arms: Wockhardt's Insulin Analogue (Recomb)
Biological: Lantus® — Basal bolus Insulin analog glargine (Lantus®) to be injected subcutaneously.
  Arms: Lantus®

SUMMARY:
This is an open label, randomized, parallel group comparison of the immunogenicity safety of Wockhardt's Recombinant Insulin Analogue with the innovator's Glargine in Type 1 diabetics patients.

DETAILED DESCRIPTION:
To evaluate and compare the Immunogenicity Safety of Wockhardt's Recombinant Insulin Analogue with innovator's Glargine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been pre-diagnosed as cases of type-1 diabetes for a period not less than 1 year
2. Male or Female Patients >= 18 and =< 55 years of age.
3. Patients with BMI of 18.0 to 30.0 kg/m2
4. Patients who are cooperative, reliable, and agree to have regular injections of insulin and are willing to comply with protocol procedures.

Exclusion Criteria:

1. A Patient who is pregnant or is currently breast-feeding.
2. A Patient with history of severe hypoglycemia within the past year
3. A Patient who is an employee of the Investigator, or a patient who has a direct involvement with the trial or other trials under the direction of the Investigator.
4. Patients who are Hepatitis B or C positive on testing or have positive medical history of HIV at screening.
5. Patients unlikely to comply with the study protocol e.g. unable to return periodically for subsequent visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in HbAlc from baseline till the end of treatment period. | 12 months

SECONDARY OUTCOMES:
Percentage change in immunogenic response. | 12 months
  Evaluating antibodies titre.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ashima Bhatia, M.D., Study Director — Wockhardt